CLINICAL TRIAL: NCT01390064
Title: Phase 1 Safety Study of a Carbohydrate Mimotope Based Vaccine With MONTANIDE ISA 51 VG Adjuvant
Brief Title: Vaccination of High Risk Breast Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110396
Record Dates: First submitted 2011-06-29; First posted 2011-07-08 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Vaccination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Initial Cohort (Experimental): Vaccination with Mimotope P10s-PADRE/MONTANIDE ISA 51 VG Subcutaneous administration 5 doses of 300 micrograms
  Interventions: Biological: Vaccination with Mimotope P10s-PADRE/MONTANIDE ISA 51 VG
- Escalation Cohort (Active Comparator): Vaccination with Mimotope P10s-PADRE/MONTANIDE ISA 51 VG Subcutaneous administration of 5 doses of 500 micrograms
  Interventions: Biological: Vaccination with Mimotope P10s-PADRE/MONTANIDE ISA 51 VG
- De-escalation Cohort (Active Comparator): Vaccination with Mimotope P10s-PADRE/MONTANIDE ISA 51 VG Subcutaneous administration of 5 doses of 100 micrograms
  Interventions: Biological: Vaccination with Mimotope P10s-PADRE/MONTANIDE ISA 51 VG

INTERVENTIONS:
Biological: Vaccination with Mimotope P10s-PADRE/MONTANIDE ISA 51 VG — All research participants will receive the Mimotope P10s-PADRE/MONTANIDE ISA 51 VG vaccine via subcutaneous (SC) injection following the schedule

SUMMARY:
Objective - Determine the safety and tolerability of a peptide mimotope-based vaccine upon immunization of breast cancer subjects.

DETAILED DESCRIPTION:
After signing Institutional Review Board (IRB) approved consent, cohorts of 3-6 stage IV breast cancer subjects will be enrolled into the study. The vaccine doses will be prepared and dispensed by the University of Arkansas for Medical Sciences (UAMS) Pharmacy following the manufacturer's instructions. Subjects will receive 1.0 mL subcutaneous (SC) injections of the vaccine on 5 separate occasions during Weeks 1, 2, 3, 7, and 19. The first cohort will begin with the 300 mg dose, and then the subsequent cohorts will escalate to 500 mg or de-escalate to 100 mg as determined by the toxicity criteria. The immunization at week 19 is considered a booster immunization. The vaccine will be administered at rotating sites on the limbs or abdomen. The study will last for approximately 12 - 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects of all races with histologically or cytologically confirmed stage IV breast cancer are eligible. The cancer may be newly diagnosed metastatic or relapsed after primary or adjunctive therapy and must not have required a treatment change for 2 months. Treatments with anti-estrogen therapy or chemotherapy are allowed. The chemotherapy regimen cannot contain steroids in the pre or post supportive care medications. If a subject is on an investigational drug, the drug must be cleared from the body over a period of 4 weeks.
* Disease staging will be done according to the American Joint Commission on Cancer (AJCC), sixth edition.
* Age 18 years and older of all races and ethnicity.
* ECOG Performance Status 0 or 1.
* Subjects must not have an active infection requiring treatment with antibiotics.
* Subjects must not have other significant medical, surgical or psychiatric conditions, or require any medication or treatment, which may interfere with compliance of the treatment regimen.
* Subjects must not have a diagnosis or evidence of organic brain syndrome, significant impairment of basal cognitive function or any psychiatric disorder that might preclude participation in the full protocol.
* Subjects must have no other current malignancies. Subjects with prior history at any time of any in situ cancer, including lobular carcinoma of the breast in situ, cervical cancer in situ, atypical melanocytic hyperplasia or Clark I melanoma in situ or basal or squamous skin cancer are eligible, provided they are disease-free at the time of registration. Subjects with other malignancies are eligible if they have been continuously disease free for ≥ 5 years prior to the time of registration.
* Subjects must not have autoimmune disorders or conditions of immunosuppression. This includes, but is not limited to being treated with corticosteroids, including oral steroids (i.e. prednisone, dexamethasone), continuous use of topical steroid creams or ointments or any steroid-containing inhalers. Subjects who have been on systemic steroids will require a 6-week washout period. Subjects who discontinue the use of these classes of medication for at least 6 weeks prior to registration are eligible if, in the judgment of the treating physician, the subject is not likely to require these classes of drugs during the treatment period. Replacement doses of steroids for subjects with adrenal insufficiency are allowed.
* Women of childbearing potential must not be pregnant (negative serum pregnancy test must be done 48 hours prior to receiving the first dose of study drug) or breastfeeding,due to the unknown effects of peptide/mimotope vaccines on a fetus or infant.
* Women of childbearing potential must be counseled to use an accepted and effective method of contraception (including abstinence) while on treatment and for a period of 18 months after completing or discontinuing treatment. Accepted methods include oral contraceptives, barrier method, Intrauterine Devices (IUDs), and abstinence.
* Subjects must have obtained a white blood cell (WBC) count ≥ 3,000/mm3 and platelet count ≥ 100,000/mm3 within 2 weeks prior to registration.
* Subjects must have a serum glutamic-oxaloacetic transaminase (SGOT)/aspartate aminotransferase test (AST) and bilirubin ≤ 2 x institutional upper limit (IUL) of normal and serum creatinine ≤ 1.8 mg/dl, all obtained within 2 weeks prior to registration.
* Subjects must be immunocompetent as measured by responsiveness to two recall antigens by skin testing.
* All subjects who wish to participate in the study must sign an informed consent approved by the UAMS Institutional Review Board (IRB).
* Laboratory tests must be completed within 2 weeks before the first dose.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Hutchins, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Initial Cohort | Escalation Cohort
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Initial Cohort | Escalation Cohort | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (17.4) | 56.0 (9.5) | 56.5 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6
Performance Status (ECOG) [Mean (Standard Deviation); unit: ECOG units on a scale 0 Best-5 Worst] | 0.0 (0.0) | 0.3 (0.6) | 0.2 (0.4)
Lines of Prior Endocrine Therapy [Mean (Standard Deviation); unit: Numbers of therapy] | 0.7 (1.2) | 1.7 (1.5) | 1.2 (1.3)
Lines of Prior Chemotherapy [Mean (Standard Deviation); unit: Numbers of therapy] | 1.3 (0.6) | 1.3 (0.6) | 1.3 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Dose-limiting Toxicity (Defined as an Adverse Event of Grade 3 or Higher)
Description: The safety and tolerability of the P10s-PADRE/MONTANIDE ISA51 VG vaccine will be determined by toxicity assessments throughout the duration of the study. Subjects will be evaluated for toxicity using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.
Time Frame: 9 weeks per subject
Measure: Number; unit: participants
Arm/Group | Initial Cohort | Escalation Cohort
Number analyzed (Participants) | 3 | 3
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 7 months during and after the vaccine was administered.
Description: All-cause Mortality AEs and Serious Adverse Events were monitored but there are none to report.
  All Other(Not Including Serious) Adverse Events have been provided in a table format.
Arm/Group | Initial Cohort | Escalation Cohort
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initial Cohort (N=3) | Escalation Cohort (N=3)
Other: Subcutaneous nodule at injection site (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) — Grade 1 - Anticipated - Definitely related to the study - Definitely related to the study Therapy
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Grade 1 - Unanticipated - Not related to the study - Not related to the study therapy
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) — Grade 1 - Unanticipated - Unlikely related to the study - Unlikely related to study therapy
Autoimmune disorder: Increase in ANA (Immune system disorders) | 1 (1) | 0 (0) — Grade 1 - Anticipated - Possibly related to study - definitely related to study therapy
Rash maculopapular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Grade 1 - Unanticipated - Definitely related to they study - Definitely related to study therapy
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Grade 1 - Unanticipated - Definitely related to they study - Possibly related to study therapy
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) — Grade 1 - Unanticipated - Not related to they study - Not related to the study therapy
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Grade 1 - Unanticipated - Not related to the study - Not related to the study therapy
Other: tender knots at the site of injections (General disorders) | 0 (0) | 1 (1) — Grade 2 - Anticipated - Definitely related to the study - Definitely related to the study therapy
Colonic hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 2- Unanticipated - Not related to the study - Not related to the study therapy
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Grade 1 - Unanticipated - Not related to the study - Not related to the study therapy
Skin induration: small lumps on abdomen at site of study drug administration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Grade 1 - Anticipated - Definitely related to the study - Not related to study therapy
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Grade 2 - Anticipated - Not related to the study - Not related to the study therapy
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Grade 2 - Unanticipated - Not related to the study - Not related to the study therapy
Skin Induration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Grade 1 - Unanticipated - Possibly related to they study - Definitely related to the study therapy
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Grade 2 - Unanticipated - Not related to the study - Not related to the study therapy
Skin induration: abdomen and right upper arm (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Grade 2 - Anticipated - Possibly related to the study - Definitely related to the study therapy
Pain of skin: constant soreness at injection sites when the area is touched (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Grade 2 - Anticipated - Possibly related to the study - Possibly related to the study therapy
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Grade 1 - Anticipated - Possibly related to the study - Possibly related to the study therapy
Other (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Grade 1 - Unanticipated - Not related to the study - Not related to the study therapy
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 (1) — Grade 1 - Unanticipated - Not related to the study - Not related to the study therapy
Other: bitten by unknown insect on the back of left leg (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Grade 2 - Unanticipated - Not related to the study - Not related to the study therapy
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) — Grade 2 - Unanticipated - Not related to the study - Not related to the study therapy
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Grade 1 - Unanticipated - Not related to the study - Not related to the study therapy
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) — Grade 1 - Unanticipated - Not related to the study - Not related to the study therapy
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Grade 2 - Unanticipated - Not related to the study - Not related to the study therapy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-11-01): https://cdn.clinicaltrials.gov/large-docs/64/NCT01390064/Prot_SAP_000.pdf